CLINICAL TRIAL: NCT02740036
Title: Quality Control of CE-Certified Phonak Hearing Aids
Brief Title: Quality Control of CE-Certified Phonak Hearing Aids - 2016_06
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Other Study IDs: Sonova2016_06
Record Dates: First submitted 2016-03-31; First posted 2016-04-15 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Hearing Aid (Successor of Phonak Audéo V90) — Successor of Phonak's Receiver-In-the-Canal (RIC) hearing aid Audéo V90.

SUMMARY:
A methodical evaluation of new CE-labelled Phonak Hearing Systems is intended to be conducted on hard of hearing participants to grant quality control prior to product launch. The aim of the investigation series is to ensure zero-defect overall performance of the new hearing systems as well as maximum benefit for the participant with the devices in comparison to previously outstanding Phonak Hearing Systems and to equivalent competitor devices.

DETAILED DESCRIPTION:
Phonak Hearing Systems pass through different development and study stages. At an early stage, feasibility studies are conducted to investigate new algorithms, features and functions in an isolated manner. If the benefit is proven, their performance is then investigated regarding interdependency between all available algorithms, features and functions running in parallel in a hearing aid (pivotal/pre-validation studies) and, as a result, they get optimized. Afterwards, and prior to product launch, the Phonak Hearing Systems undergo a final quality control in terms of clinical trials in the way as planned for this study ("phase of final inspection"). This will be a controlled, single blinded and randomised active comparator clinical evaluation which will be conducted mono centric at Sonova AG Headquarters based in Stäfa (Switzerland).

ELIGIBILITY:
Inclusion Criteria:

* Adult hearing impaired persons (minimum age: 18 years) with and without (experience with) hearing aids
* Good written and spoken (Swiss) German language skills
* Healthy outer ear
* Ability to fill in a questionnaire (p/eCRF) conscientiously
* Informed Consent as documented by signature

Exclusion Criteria:

* Contraindications to the MD in this study, e.g. known hypersensitivity or allergy to the investigational product
* Limited mobility and not in the position to attend weekly appointments in Stäfa (Switzerland)
* Limited ability to describe listening impressions/experiences and the use of the hearing aid
* Inability to produce a reliable hearing test result
* Massively limited dexterity
* Known psychological problems
* Central hearing disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2016-05; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Zero-defect performance in daily life | Four weeks
  The data, serving as primary outcomes are collected in a series of home trials taking place between the lab trial appointments. The zero-defect performance in daily life (that means: no interruptions, distortions, artefacts, feedback, system noise or other malfunctions) will be assessed with the aid of quantitative questionnaires. The results are "Yes/No" replies and open-ended.

SECONDARY OUTCOMES:
Speech intelligibility in percent in a quiet listening situation | Four weeks
  The data, serving as secondary outcomes are collected in a series of lab appointments. The speech intelligibility in quiet will be assessed with the aid of the german rhyme test "Einsilber-Reimtest nach von Wallenberg und Kollmeier" (WaKo). The result is the speech intelligibility in percent. Descriptive statistics will be executed in the form of determining the median and quartiles. Interference statistics will be executed by applying the appropriate parametric or non-parametric test, depending on the data's distribution. A significance level of 5% is pursued.
Speech intelligility in noise as signal to noise ration in dB (dB SNR) | Four weeks
  The data, serving as secondary outcomes are collected in a series of lab appointments. The speech intelligibility in noise will be assessed with the aid of the german Oldenburger sentence test. The result is the signal to noise ratio in dB (dB SNR). Descriptive statistics will be executed in the form of determining the median and quartiles. Interference statistics will be executed by applying the appropriate parametric or non-parametric test, depending on the data's distribution. A significance level of 5% is pursued.

OTHER OUTCOMES:
Initial first fit acceptance (pre-calculation) in lab | One week
  The data, serving other pre-specified outcomes are collected within the first lab appointment. The acceptance of the initial first fit will be assessed with the aid of quantitative questions within an interview. The results are points on a scale and open ended (e.g. Question: Please rate the sound quality; Answer scale: bad, poor, fair, good, excellent) . Descriptive statistics will be executed in the form of determining number of answers. Interference statistics will be executed by applying the appropriate parametric or non-parametric test, depending on the data's distribution. A significance level of 5% is pursued.
Real ear frequency responses of the hearing aids (Real Ear Measurements) | One week
  The data, serving other pre-specified outcomes are collected within the first lab appointment. The Real Ear Measurements (REMs) will be assessed with the aid of quantitative questions within an interview. The results are frequency responses (magnitude and phase of the hearing aid output as a function of frequency).

CONTACTS AND LOCATIONS:
Locations (1):
- Sonova AG, Stäfa, Canton of Zurich, Switzerland